CLINICAL TRIAL: NCT00303069
Title: A Sequential-Panel, Dose-Ranging Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Single Dose of Merck 0657nI Staphylococcus Aureus Vaccine in Healthy Adults 18 to 55 Years of Age
Brief Title: V710 First-In-Man (FIM) Study (V710-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V710-001; Formally IRB#0602011; 2010_523
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Staphylococcal Infections
Keywords: S. aureus;; Vaccine; FIM
MeSH Terms: conditions — Staphylococcal Infections | interventions — V710 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- V710 5 μg (Experimental): V710 S. aureus vaccine
  Interventions: Biological: V710
- V710 30 μg (Experimental): V710 S. aureus vaccine
  Interventions: Biological: V710
- V710 90 μg (Experimental): V710 S. aureus vaccine
  Interventions: Biological: V710
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: V710 — Single dose of V710 (at dosages of 5 μg, 30 μg, or 90 μg) intramuscularly
  Arms: V710 30 μg; V710 5 μg; V710 90 μg
Biological: Comparator: Placebo — Single dose of saline placebo intramuscularly
  Arms: Placebo

SUMMARY:
This is a randomized, Multicenter, double-blind (subject, investigator, and Merck Research Laboratories (MRL) clinical personnel directly involved in the study), placebo-controlled, dose-ranging study in healthy adults 18 to 55 years of age. It is the first in man (FIM) study evaluating the tolerability and immunogenicity of the 0657nI S. aureus vaccine. For this Phase I study, approximately 120 healthy adults will be enrolled in the study and randomized to receive a single 0.5 mL vaccination of either 0657nI S. aureus vaccine (3 different dosage levels of 5 μg, 30 μg or 90 μg of the 0657nI vaccine) or saline placebo. Vaccine/placebo will be administered intramuscularly (IM) in the deltoid muscle. Because this study will be the first study evaluating the tolerability and immunogenicity of 0657nI S. aureus vaccine in humans, a dose-escalation phase will be conducted in a small number of subjects randomized in a 3:1 ratio (n=36, consisting of 9 subjects for each of 3 vaccine dosage levels and 9 placebo subjects) to evaluate the vaccine safety at increasing dose levels of the 0657nI protein in Panel A, before expanding the enrollment to the remaining 84 subjects in Panel B.

DETAILED DESCRIPTION:
Depending on when the subject is enrolled into the study, the following will be completed: The subject will receive a single injection of SAV or placebo (an inactive substance) in the deltoid muscle of the upper arm. The subject will then be watched for 30 minutes after vaccination to monitor for allergic reactions. The subject will be asked to visit the study doctor either 6 or 9 times during the 3-month study period. Once enrolled, the subject will have blood drawn before receiving the vaccine (baseline) and up to 7 times after that at each of the required visits. The blood will be used for tests and/or for testing the subject's body's immune response to the SAV, to see if the subjects have developed immunity to S. aureus and if immunity continues up to 84 days. A Vaccination Report Card (VRC) will be provided to all participants. The participant will be asked to record oral temperatures and any reactions that occur at the SAV injection site every day for 5 days after vaccination. The participant will also be asked to record any physical adverse effects that they may experience, including headaches, nausea, muscle pain or aches, and fatigue every day for 14 days after vaccination. In additional all medications (including over the counter medications) taken during the 14 days post vaccination will be recorded and the VRC will be returned to the research staff after 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 55 years of age
* Subject is in good physical health based upon medical history, physical examination, and screening laboratory studies. NOTE: Lab studies will only be collected in Panel A, the dose-escalating portion of the study
* Subject is able to understand study procedures and agrees to participate in the study by providing written informed consent
* Subject is willing and able to participate in the entire study duration planned for 3 months (~84 days)
* Female subjects are required to have a negative urine pregnancy test immediately prior to study vaccination. Female subjects of childbearing potential must have been using an acceptable method of birth control for 2 weeks prior to enrollment, and agree to use an acceptable method of birth control for 1 month after vaccination. (Acceptable methods of birth control include use of hormonal contraceptives, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, tubal ligation, condoms, or abstinence)

Exclusion Criteria:

* Subject suffers from a chronic skin condition that predisposes the individual to the development of chronic skin or soft-tissue infections (e.g., psoriasis, chronic granulomatous disease).
* Subject developed a serious infection (e.g., bacteremia, pneumonia, mediastinitis) attributed to S. aureus in the 12 months prior to screening
* Subject has a history of anaphylaxis to aluminum-containing adjuvant or other vaccine components
* Subject has a temperature of ≥100.4ºF (≥38.0ºC), oral equivalent, within 48 hours prior to receipt of 0657nI S. aureus vaccine/placebo
* Subject has received a live virus vaccine within 30 days prior to receipt of 0657nI S. aureus vaccine/placebo or is scheduled to receive vaccination with a live virus vaccine within 30 days following study entry
* Subject has received any other licensed vaccine (including non-live virus vaccines) within 14 days prior to receipt of 0657nI S. aureus vaccine/placebo or is scheduled to receive any other licensed vaccine (including non-live virus vaccines) within 30 days following study entry. (Note: Influenza vaccines may be administered during the study, but must be given at least 7 days prior to receipt of the study vaccine or at least 15 days after receipt of the study vaccine)
* Subject was administered immunoglobulin or blood product within 90 days prior to receipt of 0657nI S. aureus vaccine/placebo or is scheduled to receive such products within 30 days following study entry
* Subject has received treatment with systemic (intramuscular, oral, or intravenous) corticosteroids or another immunosuppressive medication (e.g., calcineurin inhibitors, mycophenolate, azathioprine) in the 14 days prior to receipt of 0657nI S. aureus vaccine/placebo or is anticipated to receive such medications for a chronic medical condition during the course of the study
* Subject has a condition that requires active medical intervention or monitoring to avert serious danger to the subject's health or well-being, such as diabetes mellitus, autoimmune disease, or clinically significant chronic medical conditions that are considered progressive, including but not limited to: coronary artery disease, congestive heart failure, cardiomyopathy, progressive valvular heart disease, chronic obstructive pulmonary disease, pulmonary fibrosis, active peptic ulcer disease, chronic renal disease, chronic hepatic disease, multiple sclerosis, progressive neuropathies, or seizure disorder requiring therapy in the past 3 years
* Subject has known or suspected impairment of immunologic function including, but not limited to, the following conditions: autoimmune disease, diabetes mellitus, end-stage renal disease, hepatic insufficiency/cirrhosis, splenectomy, or HIV/AIDS
* Subject has a condition in which repeated venipuncture or injections pose more than minimal risk for the subject, such as hemophilia, other severe coagulation disorders, or significantly impaired venous access
* Subject is currently pregnant or breastfeeding, or planning to conceive within the 3-month study duration period
* Subject has clinically significant abnormalities based on the subject's medical history, physical examination, or screening laboratory studies (as described in Appendix 1 of the Multicenter protocol). NOTE: Lab studies will only be collected in Panel A, the dose escalating portion of the study
* Subject has recent history (within the past 5 years) or current evidence of drug or alcohol abuse
* Subject has a major psychiatric illness, including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, or any subject with suicidal ideation within the previous 3 years
* Subject is legally or mentally incapacitated
* Subject has participated in another clinical study in the past 4 weeks, or plans to participate in a treatment-based study or study in which an invasive procedure is to be performed while enrolled in this study. NOTE: Participation in a safety surveillance study is acceptable
* Subject has a history of any condition which, in the opinion of the investigator, may pose an additional risk for the subject or confound the results of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2005-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Harro C, Betts R, Orenstein W, Kwak EJ, Greenberg HE, Onorato MT, Hartzel J, Lipka J, DiNubile MJ, Kartsonis N. Safety and immunogenicity of a novel Staphylococcus aureus vaccine: results from the first study of the vaccine dose range in humans. Clin Vaccine Immunol. 2010 Dec;17(12):1868-74. doi: 10.1128/CVI.00356-10. Epub 2010 Oct 13. PMID 20943877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I; First Subject In: 06-Dec-2005; Last Subject Out: 31-Jul-2006. Enrollment occurred at 6 investigative sites in the United States.
Pre-assignment Details: Subject was 18 to 55 years old; in good physical health based upon medical history, physical exam, and screening tests; able to understand study procedures and provided written consent; willing and able to complete entire study; and (if female) provided negative urine pregnancy test before vaccination and using an accepted method of birth control.
Groups:
- V710 5 μg; V710 30 μg; V710 90 μg; Placebo: Panel A (dose-ranging) consisted of 36 subjects divided into 3 sequential enrollment periods (Periods 1, 2, and 3), which evaluated the safety of V710 Staphylococcus aureus vaccine at incremental dosages (5 μg, 30 μg, and 90 μg). Subjects in each period were randomized at a 3:1 ratio to receive a single intramuscular (IM) injection of either V710 (5 μg at Period 1; 30 μg in Period 2; and 90 μg in Period 3).
  Following the completion of Panel A and satisfactory interim review of the immunogenicity and safety data, the open-enrollment phase (Panel B) was initiated. Panel B consisted of 88 subjects randomized in a 1:1:1:1 ratio to receive a single IM injection of 1 of the 3 V710 dosages (5 μg, 30 μg, or 90 μg) or saline placebo. Enrollment in Panel B was stratified by age, with half of the subjects 18 to 39 years of age, the other half 40 to 55 years of age.
Period: Overall Study
Arm/Group | V710 5 μg | V710 30 μg | V710 90 μg | Placebo
Started | 31 | 28 | 34 | 31
Completed | 29 | 28 | 33 | 29
Not Completed | 2 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2
Not completed — subject moved | 1 | 0 | 0 | 0
Not completed — Recruitment into Army Reserves | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- V710 5 μg: V710 5 μg single dose at baseline.
- V710 30 μg: V710 30 μg single dose at baseline.
- V710 90 μg: V710 90 μg single dose at baseline.
- Placebo: Saline placebo single dose at baseline.
- Total: Total of all reporting groups
Arm/Group | V710 5 μg | V710 30 μg | V710 90 μg | Placebo | Total
Number analyzed (Participants) | 31 | 28 | 34 | 31 | 124
Age, Customized [Number; unit: participants]
  17 years of age and under | 0 | 0 | 0 | 0 | 0
  18 to 29 years of age | 10 | 5 | 8 | 10 | 33
  30 to 39 years of age | 7 | 8 | 12 | 5 | 32
  40 to 49 years of age | 11 | 8 | 11 | 11 | 41
  50 to 55 years of age | 3 | 7 | 3 | 5 | 18
  Over 55 years of age | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 16 | 18 | 68
  Male | 18 | 7 | 18 | 13 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 0 | 1 | 3 | 7
  Black | 9 | 8 | 4 | 4 | 25
  Hispanic-American | 1 | 1 | 2 | 0 | 4
  Multiracial | 0 | 0 | 1 | 1 | 2
  Native American | 0 | 0 | 0 | 2 | 2
  White | 18 | 19 | 26 | 21 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaccine-related Serious Adverse Experiences Following Vaccination
Description: Participants with a serious vaccine-related adverse experiences (AE) (an AE which is assessed by an investigator/qualified physician as being related to study vaccine and results in death, persistent or significant disability/incapacity, prolongs an existing inpatient hospitalization, is life-threatening, a congenital anomaly/birth defect, a cancer, or an overdose).
Time Frame: Through Day 84 postvaccination
Population: The population analyzed included all subjects who were randomized, vaccinated, and had safety follow-up.
Measure: Number; unit: Participants
Arm/Group | V710 5 μg | V710 30 μg | V710 90 μg | Placebo
Number analyzed (Participants) | 31 | 28 | 34 | 31
Participants
  Experienced a vaccine-related SAE | 0 | 0 | 0 | 0
  Did not experience a vaccine-related SAE | 31 | 28 | 34 | 31

2. Primary Outcome: Number of Participants With ≥2-fold Rise in Antibody Titer From Baseline at Day 14 Postvaccination
Time Frame: Baseline and Day 14 postvaccination
Population: The population analyzed was the per-protocol population, excluding subjects identified as protocol violators. Subjects who were found to have deviated from the protocol procedures were evaluated to determine if they should be excluded from the per-protocol analyses. These evaluations were made prior to study unblinding on a case by case basis.
Measure: Number; unit: Participants
Arm/Group | V710 5 μg | V710 30 μg | V710 90 μg | Placebo
Number analyzed (Participants) | 31 | 28 | 31 | 28
Participants
  Fold-rise in antibody titer ≥2 | 9 | 24 | 27 | 1
  Fold-rise in antibody titer <2 | 22 | 4 | 4 | 27
Statistical Analysis 1: Comparison: V710 90 μg vs Placebo; Testing was performed in a sequential manner. First, the response rate of the 90-μg group was compared to placebo and assessed for significance (using a 1-tailed α=0.025). If significant, the response rate of the 30-μg group was compared to placebo and assessed for significance. The testing continued sequentially until a non-significant result was observed or until all V710 groups had been compared with placebo; Test type: Superiority or Other; p < 0.001, Chi-squared — P-value < 0.025 considered significant; Normal approximation for testing 2 independent binomial proportions, stratified by age group (<40 yrs, ≥40 yrs); Risk Difference (RD) = 84.5, 95% CI 2-sided [65.2 to 93.6] — Risk Difference is 90 μg minus Placebo and is expressed in percentage points, confidence intervals were computed using the stratified method given by Miettinen and Nurminen
Statistical Analysis 2: Comparison: V710 30 μg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.01, Chi-squared — P-value < 0.025 considered significant; Normal approximation for testing 2 independent binomial proportions, stratified by age group (<40 yrs, ≥40 yrs); Risk Difference (RD) = 81.6, 95% CI 2-sided [61.6 to 92.0] — Risk Difference is 30 μg minus Placebo and is expressed in percentage points, confidence intervals were computed using the stratified method given by Miettinen and Nurminen
Statistical Analysis 3: Comparison: V710 5 μg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared — P-value < 0.025 considered significant; Normal approximation for testing 2 independent binomial proportions, stratified by age group (<40 yrs, ≥40 yrs); Risk Difference (RD) = 25.0, 95% CI 2-sided [6.7 to 43.8] — Risk Difference is 5 μg minus Placebo and is expressed in percentage points, confidence intervals were computed using the stratified method given by Miettinen and Nurminen

3. Secondary Outcome: Number of Participants With ≥2-fold Rise in Antibody Titer From Baseline at Day 7 Postvaccination
Time Frame: Baseline and Day 7 postvaccination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | V710 5 μg | V710 30 μg | V710 90 μg | Placebo
Number analyzed (Participants) | 31 | 28 | 33 | 30
Participants
  Fold-rise in antibody titer ≥2 | 1 | 4 | 10 | 0
  Fold-rise in antibody titer <2 | 30 | 24 | 23 | 30
Statistical Analysis 1: Comparison: V710 90 μg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared — P-value < 0.025 considered significant; Normal approximation for testing 2 independent binomial proportions, stratified by age group (<40 yrs, ≥40 yrs); Risk Difference (RD) = 30.9, 95% CI 2-sided [17.2 to 48.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: V710 30 μg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared — P-value < 0.025 considered significant; Normal approximation for testing 2 independent binomial proportions, stratified by age group (<40 yrs, ≥40 yrs); Risk Difference (RD) = 14.4, 95% CI 2-sided [1.6 to 32.1] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: V710 5 μg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared — P-value < 0.025 considered significant; Normal approximation for testing 2 independent binomial proportions, stratified by age group (<40 yrs, ≥40 yrs); Risk Difference (RD) = 3.5, 95% CI 2-sided [-8.2 to 16.9] — [estimate comment as in outcome 2, analysis 3]

ADVERSE EVENTS:
Time Frame: Following vaccination, all subjects in this study were followed for all clinical adverse experiences for 14 days postvaccination, and for vaccine-related serious adverse experiences and deaths for 84 days postvaccination (entire duration of the study).
Description: Specific systemic AEs: fatigue, headache, myalgia, and nausea for 14 days (D) postvaccination (PV). Injection-site AEs including maximum intensity/size for 5D PV. Elevated body temperatures for 5D PV. Subjects in Panel A (N=36) were actively followed for laboratory (lab) AEs for 7D PV. Any lab abnormalities at D7 PV were followed until resolution.
Arm/Group | V710 5 μg | V710 30 μg | V710 90 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/28 | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 18/31 | 19/28 | 28/34 | 17/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | V710 5 μg (N=31) | V710 30 μg (N=28) | V710 90 μg (N=34) | Placebo (N=31)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 3
Fatigue (General disorders) | 5 | 3 | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0
Injection-site erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3
Injection-site pain (Skin and subcutaneous tissue disorders) | 14 | 17 | 20 | 7
Injection-site swelling (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 0/11 | 0/9 | 2/9 | 0/7
Blood bilirubin increased (Investigations) | 0/11 | 0/9 | 1/9 | 0/7
Hemoglobin decreased (Investigations) | 1/11 | 0/9 | 1/9 | 0/7
Protein urine present (Investigations) | 1/11 | 0/9 | 0/9 | 1/7
White blood cell count decreased (Investigations) | 0/11 | 0/9 | 1/9 | 0/7
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 7
Headache (Nervous system disorders) | 6 | 7 | 6 | 4
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.